CLINICAL TRIAL: NCT07218991
Title: Wearable Echolocation Aids Using Parametric Sound
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 24-0032
Record Dates: First submitted 2025-02-11; First posted 2025-10-21 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Low Vision
Keywords: low vision; visual impairment; blindness; blind; visual aid; visual rehabilitation; sensory compensation; echolocation; parametric sound; parametric sound technology; wearable echolocation device; echolocation technology; directional sound waves; echolocation headphones; assistive device; echolocation skills; ultrasound waves; sound waves; adaptive low vision navigation aid; low vision simulation goggles; navigation aid; low vision simulator
MeSH Terms: conditions — Vision, Low; Vision Disorders; Blindness; Echolocation

STUDY DESIGN:
Intervention Model Description: Subjects will be divided into two groups who will both perform identical study activities, performing a trial with the study device and another without the study device, however, in a different order.
Who Masked: Outcomes Assessor
Masking Description: Subjects will be randomly assigned to one of two groups. Both groups will perform identical study activities, though the order of activities will be different. Group assignment will not be provided to the outcomes assessor so as to avoid influencing the analysis of the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Wearing a Low-Vision Simulator without the Wearable Echolocation Device (No Intervention): The participant will be wearing a low-vision simulator and navigating a pathway randomly populated with obstacles. They will then perform the same trial, wearing the low vision simulator, navigating the same pathway with obstacles randomly rearranged; however, the participants will use the Wearable Echolocation Device to assist with navigation.
- Group 2- Wearing a Low-Vision Simulator with the Wearable Echolocation Device (Active Comparator): The participants will be wearing the low-vision simulator and the wearable echolocation Device for the first test to assist with navigating the pathway randomly populated with obstacles. The participant will then perform the same test, wearing the low-vision simulator without the Wearable Echolocation Device, navigating the same pathway with randomly rearranged obstacles.
  Interventions: Device: Wearable Echolocation Device

INTERVENTIONS:
Device: Wearable Echolocation Device — The device features many parametric speakers housed in a plastic case. The parametric speakers emit directional sound waves that return to the source with varying wavelengths depending on the distance of the surrounding objects. The device is designed to be worn by the subject either using a lanyard on the subject's neck, or on the subject's wrist.
  Arms: Group 2- Wearing a Low-Vision Simulator with the Wearable Echolocation Device

SUMMARY:
The objective of this study is to study a novel device designed to aid patients with impaired vision to safely navigate their environment. Subjects for this study will be individuals with normal vision, either with or without correction. The subjects will wear a device to simulate impaired vision and will be asked to walk a path with randomly placed obstacles during two trials. One of the trials will consist of the subject wearing the simulator alone. The other trial will consist of the subject wearing the simulator and the study device. The study device is designed to be worn by the study subject and will emit tones to indicate obstacles in the environment as the subject walks on the path with random obstacles. The tones will indicate that there is an obstacle in the individual's path and will increase in intensity as the subject moves closer to the object.Invest

DETAILED DESCRIPTION:
The objective of this project is to study visually impaired individuals' ability to develop echolocation skills using simple, wearable, echolocation devices that will not be cost prohibitive to most Americans and that would allow for greater availability to the visually impaired community. These echolocation devices emit parametric sound, a directional beam of ultrasound waves that interact with sound waves and surrounding objects, through goggles, watches, lanyards or even walking canes. This allows the visually impaired individual to detect sound waves as they reflect off their surroundings and return to the patient's ears in unique patterns resembling their external environment. This device would enable individuals to create a raw mental image of their surroundings and any obstacles along their path.

The primary endpoint for this pilot study is to assess the feasibility of such echolocation devices as an adaptive low vision navigation aid on healthy subjects using low vision simulation goggles. Several metrics will be observed and recorded to measure how well echolocation technology addresses challenges associated with visual impairment and downstream factors. These metrics will include gait initiation, termination analysis via the Zeno-Walkway system, electromyography (EMG) of key muscles involved in gait termination, participant preference of echolocation wearable device modularity, and general survey questions.

The secondary study endpoint is to implement the use of echolocation technology among members of the blind or visually impaired population as a clinical aid and study the impact that this technology has on their quality of life and added downstream health implications longitudinally.

A final objective of this study is to seek feedback, not only on the use of any echolocation device to navigate but, to obtain feedback on subjects' experience with the specific study device, the Wearable Echolocation Device.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent in a manner approved by the Institutional Review Board (IRB) and is willing and able to comply with the trial procedures.
* Adults at least 18 years of age and no older than 100 years of age at the time of consent.
* Individuals in good health who can perform daily activities without assistance and can walk independently.
* Normal vision (with or without corrective lenses) if there is no uncorrectable visual impairment.

Exclusion Criteria:

* History of gait problems.
* Foot or leg impairments.
* Hearing impairment.
* Vertigo or other balance problems.
* Pregnant individuals.
* Any medical condition that, in the opinion of the investigator, would place the subject at increased risk for participation.
* Medications that may cause dizziness or weakness.
* Concurrent participation on another research study.
* Use of an investigational agent in the 30 days prior to signing informed consent.
* History of prior non-compliance.
* Presence or history of psychiatric condition (including anxiety, psychosis, drug, or alcohol addiction) that would, in the opinion of the investigator, make it difficult for the subject to comply with the study procedures or follow the investigators instructions.
* Non-English-speaking individuals.
* Individuals from special or vulnerable populations (i.e., adults unable to consent, minors, incarcerated individuals).
* Body weight greater than 700 pounds.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2027-06-14 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Stride Length for Visually Impaired Individuals with Implementation of Echolocation Technology | Baseline (pre-training) and immediately post-training (same 30 minute session)
  Stride length will be measured using the Zeno Walkway system, an electronic, pressure-sensitive mat connected to a PC that automates the measurement of spatial and temporal aspects of gait. The walkway's high-resolution sensors capture real-time data as participants walk across it. Each participant will walk on the instrumented mat for approximately 30 minutes, allowing for detailed analysis of stride length. Mean stride length (in meters) will be calculated from multiple trials to assess changes following implementation of echolocation technology.
Change in Cadence for Visually Impaired Individuals with Implementation of Echolocation Technology | Baseline (pre-training) and immediately post-training (same 30 minute session)
  Cadence (steps per minute) will be assessed using the Zeno Walkway system, an electronic, pressure-sensitive mat that captures real-time gait data. Participants will walk across the instrumented walkway for approximately 30 minutes. The system will automatically record and calculate the average number of steps per minute to evaluate changes in cadence following implementation of echolocation technology.
Change in Walking Velocity for Visually Impaired Individuals with Implementation of Echolocation Technology | Baseline (pre-training) and immediately post-training (same 30 minute session)
  Walking velocity will be measured using the Zeno Walkway system, an electronic, pressure-sensitive mat that captures spatial and temporal aspects of gait. Participants will walk across the walkway for approximately 30 minutes. The system will automatically calculate average walking velocity (in meters per second) based on distance and time. This outcome will be used to evaluate improvements in gait speed following implementation of echolocation technology.
Change in Body Mass Index (BMI) for Visually Impaired Individuals with Implementation of Echolocation Technology | Baseline (pre-training) and immediately post-training (same 30 minute session)
  Body Mass Index (BMI) will be calculated using standard anthropometric measures of height and weight (weight in kilograms divided by height in meters squared). Measurements will be taken at each study visit to assess any change in BMI that may occur following implementation of echolocation technology.

OTHER OUTCOMES:
Participant-Reported Experience with Echolocation Device | Day 1
  Participants will complete the "Wearable Echolocation Aids Using Parametric Sound: Post-Trials Survey" to evaluate their experience using the echolocation device during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Praveena M Gupta, PhD OD FAAO, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2019 Blindness and Vision Impairment Collaborators; Vision Loss Expert Group of the Global Burden of Disease Study. Trends in prevalence of blindness and distance and near vision impairment over 30 years: an analysis for the Global Burden of Disease Study. Lancet Glob Health. 2021 Feb;9(2):e130-e143. doi: 10.1016/S2214-109X(20)30425-3. Epub 2020 Dec 1. PMID 33275950
- [Background] Varadaraj V, Ehrlich JR, Swenor BK. Vision Impairment Has Implications for Aging and Health Outcomes, Beyond Ophthalmology. JAMA Netw Open. 2022 May 2;5(5):e2214610. doi: 10.1001/jamanetworkopen.2022.14610. No abstract available. PMID 35608864
- [Background] Ong SR, Crowston JG, Loprinzi PD, Ramulu PY. Physical activity, visual impairment, and eye disease. Eye (Lond). 2018 Aug;32(8):1296-1303. doi: 10.1038/s41433-018-0081-8. Epub 2018 Apr 3. PMID 29610523
- [Background] Thaler L, Goodale MA. Echolocation in humans: an overview. Wiley Interdiscip Rev Cogn Sci. 2016 Nov;7(6):382-393. doi: 10.1002/wcs.1408. Epub 2016 Aug 19. PMID 27538733
- [Background] Swenor BK, Ehrlich JR. Ageing and vision loss: looking to the future. Lancet Glob Health. 2021 Apr;9(4):e385-e386. doi: 10.1016/S2214-109X(21)00031-0. Epub 2021 Feb 16. No abstract available. PMID 33607013
- [Background] Sohl-Dickstein J, Teng S, Gaub BM, Rodgers CC, Li C, DeWeese MR, Harper NS. A Device for Human Ultrasonic Echolocation. IEEE Trans Biomed Eng. 2015 Jun;62(6):1526-1534. doi: 10.1109/TBME.2015.2393371. Epub 2015 Jan 16. PMID 25608301
- [Background] Norman LJ, Dodsworth C, Foresteire D, Thaler L. Human click-based echolocation: Effects of blindness and age, and real-life implications in a 10-week training program. PLoS One. 2021 Jun 2;16(6):e0252330. doi: 10.1371/journal.pone.0252330. eCollection 2021. PMID 34077457
- See also: Echolocation Headphones — https://doi.org/10.1007/s00146-017-0766-8
- See also: Approaches to Reduce Vision Impairment and Promote Eye Health — https://www.ncbi.nlm.nih.gov/books/NBK402367/
- See also: Echolocation Headphones — http://aisencaro.com/echo.html